CLINICAL TRIAL: NCT04980963
Title: Cognitive Support Technology for Postsecondary Students With Autism Spectrum Disorder: A Randomized Clinical Trial at the Intervention Efficacy Stage of Research
Brief Title: Cognitive Support Technology for Postsecondary Students With Autism Spectrum Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kent State University (Other)
Collaborators: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20-069
Record Dates: First submitted 2020-09-17; First posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: A minimum total of 90 students will be recruited for the study. Study personnel will recruit 30 students in each of years 2, 3, and 4. Of the 30 students per year, 15 will be randomly assigned to the full treatment intervention and 15 students will be randomly assigned to the control group. Participants will range in age from approximately 18 years to 25 years, but all ages are welcome to participate.
  The selection of the target population for this research study is based on the bleak employment outcomes of students with ASD compared to students without disabilities. In addition, it is based on the lack of practices that integrate the cognitive and vocational needs of students with ASD who are pursuing postsecondary education to help them successfully complete academic requirements, address career development, enhance career readiness skills, and obtain and maintain employment.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full Treatment (Experimental): Steps of the Intervention Condition. Following an in-person session in which a pretest assessment is completed, each member of the intervention group will participate in three face-to-face sessions with the interventionist at the student's campus or at the interventionist's office to complete the CST component of the intervention. Taking into consideration available psychoeducational assessment data, functional assessments from other agencies, and the participant's self-report regarding the functional difficulties that result from his or her ASD-related cognitive impairments, Scherer's (2012) Matching Person and Technology (MPT) protocol will guide the CST assessment. For purposes of the CST component of this intervention, the technological platform for cognitive accommodations will be an iPad II that is provided to each intervention-group participant at no charge (including wireless access if needed). The interventionist will provide training in the use of the iPad if necessary.
  Interventions: Behavioral: Cognitive Support Technology (CST)
- Abbreviated Treatment (Active Comparator): Steps of the Control Condition. Following an in-person session in which the pretest assessment is completed, each member of the control group will participate in two telephone or Skype sessions with the interventionist to discuss her or his needs for electronic cognitive supports. An abbreviated version of Scherer's (2012) MPT assessment will be administered via telephone or Skype in the first of these virtually-administered sessions. In the second telephone or Skype session, the interventionist will summarize the results of the abbreviated MPT assessment, suggest a variety of cognitive enhancement apps for tablet computers or smart phones that the control group participant can consider.
  Interventions: Behavioral: Cognitive Support Technology (CST)

INTERVENTIONS:
Behavioral: Cognitive Support Technology (CST) — Cognitive Support Technology (CST) products and strategies are used to help people with disabilities compensate for or accommodate cognitive limitations (including those related to interpersonal communication and social cognition) that present difficulties for them in the performance of desired social roles, especially education and employment. CSTs may be mainstream everyday technologies such as tablet computers or they may be specialized devices designed for specific goals such as step-by-step instruction in the performance of a particular task (Scherer, 2012).

SUMMARY:
This study will fill important knowledge gaps in the availability of best practices that use innovative methods to integrate the cognitive and vocational needs of students with Autism Spectrum Disorder (ASD) who will be transitioning from 2- and 4-year postsecondary education to employment. Best practices exist from the assistive technology (AT) field to help people compensate for cognitive impairments, and from the vocational rehabilitation (VR) field to enhance employment outcomes for individuals with disabilities. However, these practices have not been integrated to provide needed supports and services to improve the employment outcomes of students with ASD. The study's goal is to expand the availability of innovative practices by testing the efficacy of a technology-driven, long-term, and resource-rich individualized support program that merges assistive technology for cognition and vocational rehabilitation practices. The end products will include technology application guidelines, training and procedural manuals, and resource information that rehabilitation professionals and students with ADS can utilize to enhance technology and mentoring proficiency, academic success, self-determination, and long-term career success for students with ASD.

The knowledge to be gained from this research will have a beneficial impact on students with ASD, rehabilitation professionals, higher education personnel, case managers, and employers who work with people with ASD. There is strong potential for the students to develop skills that will help them succeed in learning as well as employment settings. The ultimate benefit of research activities for the target population will be seen in the improved capacity for postsecondary students with ADS to utilize state-of-the-art technology to accommodate disability-related limitations, address career readiness, and to prepare for and obtain employment after graduation.

Because the risks to subjects are no greater than those associated with everyday life and because the study staff will refer students who are in psychological distress or medical emergency situations to appropriate resources in the community, the minimal risks of this study justify the considerable benefits that this study will yield. Not only will the study benefit participating students, it stands to make important contributions to the knowledge bases in the fields of assistive technology and rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Must be a post-secondary student enrolled in degree programs at two-year and four-year colleges or universities within a 60-mile radius of Kent, Ohio
* Must have a clinical diagnosis of Autism Spectrum Disorder

Exclusion Criteria:

* No other exclusion criteria will be applied

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Grade Point Average (GPA) | Baseline (enrollment in study), 6 months, and 1 year (study completion)
  Participant GPA

SECONDARY OUTCOMES:
Current academic standing | Baseline (enrollment in study), 6 months, and 1 year (study completion)
Post-Secondary Enrollment Status | Baseline (enrollment in study), 6 months, and 1 year (study completion)
  % of participants still enrolled in a postsecondary program
Satisfaction with current living status and transportation access | Baseline (enrollment in study), 6 months, and 1 year (study completion)
  Measured using single item 5-point Likert question on questionnaire
Satisfaction with Social Support | Baseline (enrollment in study), 6 months, and 1 year (study completion)
  Measured using single item 5-point Likert question on questionnaire
Current Employment Status | Baseline (enrollment in study), 6 months, and 1 year (study completion)
  Three items on questionnaire including dichotomous employment question (e.g., are you employed?), if yes, number of hours employed and weekly earnings.
% of Participants Receiving Disability Benefits | Baseline (enrollment in study), 6 months, and 1 year (study completion)
  Whether participants receive SSDI and/or SSI benefits or not
Depression Symptoms | Baseline (enrollment in study), 6 months, and 1 year (study completion)
  Measured using Beck Depression Inventory- II (BDI-II)
Overall Health Status | Baseline (enrollment in study), 6 months, and 1 year (study completion)
  Measured using RAND 36-item Health Survey
Perceived Stress | Baseline (enrollment in study), 6 months, and 1 year (study completion)
  Measured using Perceived Stress Scale- 10
Acceptance of Disability | Baseline (enrollment in study), 6 months, and 1 year (study completion)
  Measured using the Acceptance of Disability Scale- Short Form
Quality of Life (QoL) | Baseline (enrollment in study), 6 months, and 1 year (study completion)
  Measured using the Qualify of Life Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Kent State University, Kent, Ohio, United States

IPD SHARING:
Plan to Share IPD: No